CLINICAL TRIAL: NCT02600520
Title: 1.2% Rosuvastatin Versus 1.2% Atorvastatin Local Drug Delivery in Treatment of Intrabony Defects in Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Rosuvastatin With Atorvastatin in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor & Head, Department of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014X
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rosuvastatin Group (Active Comparator): SRP followed by RSV gel LDD
  Interventions: Drug: SRP with RSV gel LDD
- Atorvastatin Group (Active Comparator): SRP followed by ATV gel LDD
  Interventions: Drug: SRP with ATV gel LDD
- Placebo group (Placebo Comparator): SRP followed by placebo gel LDD
  Interventions: Drug: SRP with placebo gel LDD

INTERVENTIONS:
Drug: SRP with RSV gel LDD — After SRP, 1.2% Rosuvastatin (RSV) gel was delivered subgingivally into the pocket
  Arms: Rosuvastatin Group
Drug: SRP with ATV gel LDD — After SRP, 1.2% Atorvastatin (ATV) gel was delivered subgingivally into the pocket
  Arms: Atorvastatin Group
Drug: SRP with placebo gel LDD — After SRP, placebo gel was delivered subgingivally into the pocket
  Arms: Placebo group

SUMMARY:
The present study is designed as a single-centre, randomized, controlled clinical trial to evaluate and compare the clinical and radiographic efficacy of two local drug delivery systems containing 1.2% RSV gel and 1.2% ATV gel in treatment of intrabony defects in patients with chronic periodontitis as an adjunct to SRP.

DETAILED DESCRIPTION:
Background: Rosuvastatin (RSV) and Atorvastatin (ATV) are known to inhibit osteoclastic bone resorption and were proposed to have osteostimulative properties by causing osteoblast differentiation in vivo and in vitro as shown by an increase in matrix formation. The aim of the present study is to evaluate and compare the efficacy of 1.2% RSV and 1.2% ATV gel as local drug delivery systems in adjunct to scaling and root planning (SRP) for the treatment of intrabony defects in patients with chronic periodontitis (CP).

Methods: A total of 90 intrabony defects were treated with either 1.2% RSV, 1.2% ATV or placebo gel LDD after SRP. Clinical parameters (plaque index, modified sulcus bleeding index, probing depth and clinical attachment level) were recorded at baseline and 6 months. Radiographic intrabony defect depth change was calculated on standardized radiographs by using image analysis software at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with PD ≥5mm or CA loss ≥4mm and vertical bone loss ≥3 mm on intraoral periapical radiographs with no history of periodontal therapy or use of antibiotics in the preceding 6 months were included

Exclusion Criteria:

* Patients with a known systemic disease;
* known or suspected allergy to statin group;
* on systemic statin therapy;
* with aggressive periodontitis;
* who used tobacco in any form;
* alcoholics;
* immunocompromised patients;
* pregnant or lactating females were excluded from the study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in intrabony defect depth from baseline to 6 months | Baseline to 6 months
  Radiographic defect depth reduction (DDR) in the baseline to 6 months interval wiil be measured

SECONDARY OUTCOMES:
Change in plaque index (PI) from baseline to 6 months | Baseline to 6 months
  Reduction in plaque index (PI) from baseline to 6 months wiil be measured
Change in modified sulcus bleeding index (mSBI) from baseline to 6 months | Baseline to 6 months
  Reduction in modified sulcus bleeding index (mSBI) from baseline to 6 months wiil be measured
Change in probing depth (PD) from baseline to 6 months | Baseline to 6 months
  Reduction in probing depth (PD) from baseline to 6 months wiil be measured
Change in clinical attachment (CA) level from baseline to 6 months | Baseline to 6 months
  Reduction in clinical attachment (CA) level from baseline to 6 months wiil be measured